CLINICAL TRIAL: NCT06186700
Title: Effect of Pentoxifylline on Preventing Chemotherapy-induced Toxicities in Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Omar Hamdy, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-147-2
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Female; Breast Cancer Patients; Neoadjuvant Therapy; Doxorubicin; Taxane-induced Peripheral Neuropathy
Keywords: neoadjuvant chemotherapy, pentoxiphyllin, doxorubicin, cyclophosphamide, mucositis, quality of life
MeSH Terms: conditions — Mucositis | interventions — Pentoxifylline; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentoxifylline group (Active Comparator): The patient will take 400 mg tablets of Pentoxifylline, 3 tablets per day, starting from the first day of the first cycle of doxorubicin/cyclophosphamide till finishing the cycles of neoadjuvant chemotherapy comprised intravenous Doxorubicin 60 mg/m²/cycle with intravenous Cyclophosphamide 600 mg/m²/cycle for four cycles, followed by weekly paclitaxel, dose-dense paclitaxel or docetaxel.
  Interventions: Drug: Pentoxifylline 400mg plus chemotherapy
- Control group (Other): The patient will take standard neoadjuvant chemotherapy, including doxorubicin/cyclophosphamide, followed by a taxane regimen as per the medical committee.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Pentoxifylline 400mg plus chemotherapy — The patient will take 400 mg tablets of Pentoxifylline, 3 tablets per day, starting from the first day of the first cycle of doxorubicin/cyclophosphamide till finishing the cycles of neoadjuvant chemotherapy comprised intravenous Doxorubicin 60 mg/m²/cycle with intravenous cyclophosphamide 600 mg/m²/cycle for four cycles, followed by weekly paclitaxel, dose-dense paclitaxel or docetaxel.
  Other Names: Intravenous doxorubicin; Intravenous cyclophosphamide; Intravenous taxane; oral pentoxifylline
  Arms: Pentoxifylline group
Drug: Chemotherapy — The patient will take chemotherapy cycle comprised intravenous Doxorubicin 60 mg/m²/cycle with intravenous Cyclophosphamide 600 mg/m²/cycle for four cycles, followed by weekly paclitaxel, dose-dense paclitaxel or docetaxel..
  Arms: Control group

SUMMARY:
This clinical trial is a randomized clinical trial that aims to assess the usefulness of adding pentoxifylline to the neoadjuvant chemotherapy treatment protocol of doxorubicin/cyclophosphamide fllowed by taxane for breast cancer patients to decrease the incidence of developing toxicities, and enhance the quality of patient life using the EQ-5D-3L questionnaire. The participant will administer Pentoxifylline oral tablets three times per day along with the treatment protocol, starting from the first doxorubicin/cyclophosphamide cycle till the end of the chemotherapy cycles. The researchers will compare the incidence and grade of mucosities, neuropathy, and other chemotherapy-related toxicities in the presence or absence of oral pentoxifylline.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients >18 years old with histologic confirmation of invasive breast cancer
2. Planned to administer neoadjuvant chemotherapy protocol comprised of doxorubicin/ cyclophosphamide followed by paclitaxel (AC/T)
3. Adequate hepatic, renal, and bone marrow functions

Exclusion Criteria:

1. Patients on a treatment regimen of phosphodiesterase inhibitors
2. Patients who are taking antiplatelet or anticoagulant treatment
3. Patients who are allergic to phosphodiesterase inhibitors
4. History of recent hemorrhagic events
5. Active peptic ulcer
6. patients who have mouth or teeth problem.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
The incidence of grade 2 or more peripheral neuropathy in the two groups using Common Terminology Criteria Adverse Event grading | 6 months
  The number of patients reported grade 2 or more peripheral neuropathy in the two groups.

SECONDARY OUTCOMES:
The incidence of grade 2 or more oral mucositis in the two groups using Common Terminology Criteria Adverse Event grading | 6 months
  The number of patients who reported grade 2 or more oral mucositis adverse effects during the treatment period
The incidence of grade 2 or more anemia in the two groups using Common Terminology Criteria Adverse Event grading | 6 months
The incidence of grade 2 or more febrile neutropenia in the two groups using Common Terminology Criteria Adverse Event grading | 6 months
the incidence of gastrointestinal side effects including: abdominal discomfort, bloating, diarrhea, constipation will be assessed in the two groups using Common Terminology Criteria Adverse Event grading | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Center of Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Dewidar SA, Mansour NO, Hamdy O, Eltantawy A, Soliman MM, Shams MEE. Assessing the efficacy and safety of pentoxifylline in preventing chemotherapy-induced peripheral neuropathy and mucositis in breast cancer patients. Front Pharmacol. 2025 Oct 14;16:1678161. doi: 10.3389/fphar.2025.1678161. eCollection 2025. PMID 41164763